CLINICAL TRIAL: NCT03000101
Title: New Insight and Knowledge on Anti-inflammatory Effectiveness of Dietary Phenolics (NIKE)
Brief Title: Study of the Role of Pomegranate Juice Ellagitannins in the Modulation of Inflammation in Inflammatory Bowel Disease
Acronym: POME2016
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other); Conserve Italia (Unknown); GAT Foods (Other)
Responsible Party: Principal Investigator, andrea belluzzi, MD phD, Andrea Belluzzi, MD PhD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RBSI14LHMB; SIR Programme no. RBSI14LHMB (Other Grant/Funding Number: MIUR Italian Ministry of Education, University and Research)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Biomarkers; Colitis; Colitis, Ulcerative; Colonic Diseases; Crohn Disease; Digestive System Diseases; Fruit; Fruit and Vegetable Juices; Gastroenteritis; Gastrointestinal Diseases; Humans; Hydrolysable Tannins; Inflammation; Inflammatory Bowel Disease; Intestinal Diseases; Punicaceae
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Colitis; Colonic Diseases; Digestive System Diseases; Gastroenteritis; Gastrointestinal Diseases; Inflammation; Inflammatory Bowel Diseases; Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate juice (Experimental): The pomegranate juice is 100% pomegranate juice, not from concentrate.
  Interventions: Other: 100% pomegranate juice
- Placebo beverage (Placebo Comparator): The placebo beverage consists in water added with sugar and citric acid.
  Interventions: Other: placebo beverage

INTERVENTIONS:
Other: 100% pomegranate juice — 125 mL of 100% pomegranate juice twice daily for 12 weeks
  Arms: Pomegranate juice
Other: placebo beverage — 125 mL of placebo beverage twice daily for 12 weeks
  Arms: Placebo beverage

SUMMARY:
The aim of this research is to study the effects of a pomegranate juice on calprotectin levels in patients suffering of inflammatory bowel disease (IBD) in clinical remission. Fecal calprotectin levels, surrogate marker of mucosal inflammation, will be measured from baseline to 12 weeks later (end of intervention). Systemic and mucosal changes of biochemical and molecular inflammatory response markers will be also assessed.

DETAILED DESCRIPTION:
The main purpose of the intervention trial is to assess the possible effect of pomegranate juice consumption on reducing fecal calprotectin (FC) levels in volunteers suffering from IBD with a high risk of clinical relapse. In detail, the objectives of this intervention are as follows: (i) assessing the changes in FC levels in the two groups (active treatment, control) from baseline to 12 weeks later (primary outcome); (ii) investigating the systemic and mucosal modifications of selected biochemical and molecular inflammatory response markers in the two groups after 12 weeks of the intervention compared with baseline (secondary outcomes); (iii) evaluating circulating and urinary ellagitannin-derived metabolites from regular pomegranate juice consumption in the two groups before and after the intervention.

The detailed study protocol is published in the Trials journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ulcerative Colitis (diagnosed on the base of clinic, endoscopic, and histologic criteria) in clinical remission (SCCAI = 0) from at least three months and in stable therapy (without therapeutic modifications in the three previous months) with mesalazine, immunomodulators and/or biologics.
* Patients affected by Crohn's Disease, particularly involving sigmoid colon and rectum (diagnosed on the base of clinic, endoscopic, and histologic criteria) in clinical remission (CDAI < 150) from at least three months and in stable therapy (without therapeutic modifications in the three previous months) with mesalazine A, immunomodulators and/or biologics.
* Fecal calprotectin at baseline ≥ 100 microg/g.
* Signed informed consent.

Exclusion Criteria:

* Patients affected by Ulcerative Colitis and Crohn's Disease with severe endoscopic disease activity (Ulcerative Colitis: Mayo Endoscopic Score = 3; Crohn's Disease: Simple Endoscopic Score SES-CD > 15).
* Patients on steroid therapy in the two previous months.
* Patients in therapy with warfarin or other anticoagulants.
* Known or supposed hypersensitivity to fruit and/or juice of pomegranate.
* Women in fertile age which refuse to use contraceptives specified in the study (oral contraception, IUD) and breastfeed women.
* Diabetic patients and other patients with severe clinical conditions which the investigator consider to contraindicate patient participation at the study.
* Therapy modifications and/or assumption of experimental therapies within three months before the study inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Changes in fecal calprotectin | Baseline and 12 weeks
  Change from baseline in fecal neutrophil-derived protein calprotectin, surrogate marker of mucosal improvement, after 12 weeks of consumption of experimental or placebo beverage, in subjects affected by IBD in clinical remission.

SECONDARY OUTCOMES:
Changes in plasma concentration of ellagitannin metabolites | Baseline and 12 weeks
  Change from baseline in plasma concentration of ellagitannin metabolites after 12 weeks of intervention.
Changes in circulating cytokines levels | Baseline and 12 weeks
  Change from baseline in plasma levels of cytokines after 12 weeks of intervention.
Changes in circulating trimethylamine-N-oxide (TMAO) levels | Baseline and 12 weeks
  Change from baseline in plasma levels of TMAO after 12 weeks of intervention.
Changes in gene expression levels in peripheral blood mononuclear cells (PBMC) | Baseline and 12 weeks
  Change from baseline in expression levels of selected genes in PBMC by qPCR after 12 weeks of intervention.
Changes in gene expression levels in intestinal biopsies | Baseline and 12 weeks
  Change from baseline in expression levels of selected genes in intestinal biopsies by qPCR after 12 weeks of intervention.
Changes in urinary ellagitannin metabolite excretion | Baseline and 12 weeks
  Change from baseline in urinary ellagitannin metabolite excretion after 12 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Danesi, PhD, Study Director — Department of Agri-Food Sciences and Technologies, University of Bologna; Luigi Ricciardiello, MD, Prof, Principal Investigator — Department of Medical and Surgical Sciences, University of Bologna
Locations (1):
- U.O. Gastroenterologia - Azienda Ospedaliero-Universitaria di Bologna, Policlinico Sant'Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Best WR, Becktel JM, Singleton JW. Rederived values of the eight coefficients of the Crohn's Disease Activity Index (CDAI). Gastroenterology. 1979 Oct;77(4 Pt 2):843-6. PMID 467941
- [Background] Biasi F, Astegiano M, Maina M, Leonarduzzi G, Poli G. Polyphenol supplementation as a complementary medicinal approach to treating inflammatory bowel disease. Curr Med Chem. 2011;18(31):4851-65. doi: 10.2174/092986711797535263. PMID 21919842
- [Background] Costa F, Mumolo MG, Ceccarelli L, Bellini M, Romano MR, Sterpi C, Ricchiuti A, Marchi S, Bottai M. Calprotectin is a stronger predictive marker of relapse in ulcerative colitis than in Crohn's disease. Gut. 2005 Mar;54(3):364-8. doi: 10.1136/gut.2004.043406. PMID 15710984
- [Background] D'Inca R, Dal Pont E, Di Leo V, Ferronato A, Fries W, Vettorato MG, Martines D, Sturniolo GC. Calprotectin and lactoferrin in the assessment of intestinal inflammation and organic disease. Int J Colorectal Dis. 2007 Apr;22(4):429-37. doi: 10.1007/s00384-006-0159-9. Epub 2006 Jul 13. PMID 16838143
- [Background] D'Amore S, Vacca M, Graziano G, D'Orazio A, Cariello M, Martelli N, Di Tullio G, Salvia R, Grandaliano G, Belfiore A, Pellegrini F, Palasciano G, Moschetta A. Nuclear receptors expression chart in peripheral blood mononuclear cells identifies patients with Metabolic Syndrome. Biochim Biophys Acta. 2013 Dec;1832(12):2289-301. doi: 10.1016/j.bbadis.2013.09.006. Epub 2013 Sep 21. PMID 24060638
- [Background] Daperno M, D'Haens G, Van Assche G, Baert F, Bulois P, Maunoury V, Sostegni R, Rocca R, Pera A, Gevers A, Mary JY, Colombel JF, Rutgeerts P. Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD. Gastrointest Endosc. 2004 Oct;60(4):505-12. doi: 10.1016/s0016-5107(04)01878-4. PMID 15472670
- [Background] D'Haens G, Ferrante M, Vermeire S, Baert F, Noman M, Moortgat L, Geens P, Iwens D, Aerden I, Van Assche G, Van Olmen G, Rutgeerts P. Fecal calprotectin is a surrogate marker for endoscopic lesions in inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2218-24. doi: 10.1002/ibd.22917. Epub 2012 Feb 16. PMID 22344983
- [Background] Espin JC, Gonzalez-Barrio R, Cerda B, Lopez-Bote C, Rey AI, Tomas-Barberan FA. Iberian pig as a model to clarify obscure points in the bioavailability and metabolism of ellagitannins in humans. J Agric Food Chem. 2007 Dec 12;55(25):10476-85. doi: 10.1021/jf0723864. Epub 2007 Nov 9. PMID 17990850
- [Background] Foell D, Frosch M, Sorg C, Roth J. Phagocyte-specific calcium-binding S100 proteins as clinical laboratory markers of inflammation. Clin Chim Acta. 2004 Jun;344(1-2):37-51. doi: 10.1016/j.cccn.2004.02.023. PMID 15149869
- [Background] Geboes K, Riddell R, Ost A, Jensfelt B, Persson T, Lofberg R. A reproducible grading scale for histological assessment of inflammation in ulcerative colitis. Gut. 2000 Sep;47(3):404-9. doi: 10.1136/gut.47.3.404. PMID 10940279
- [Background] Gimenez-Bastida JA, Larrosa M, Gonzalez-Sarrias A, Tomas-Barberan F, Espin JC, Garcia-Conesa MT. Intestinal ellagitannin metabolites ameliorate cytokine-induced inflammation and associated molecular markers in human colon fibroblasts. J Agric Food Chem. 2012 Sep 12;60(36):8866-76. doi: 10.1021/jf300290f. Epub 2012 Apr 16. PMID 22463485
- [Background] Larrosa M, Gonzalez-Sarrias A, Yanez-Gascon MJ, Selma MV, Azorin-Ortuno M, Toti S, Tomas-Barberan F, Dolara P, Espin JC. Anti-inflammatory properties of a pomegranate extract and its metabolite urolithin-A in a colitis rat model and the effect of colon inflammation on phenolic metabolism. J Nutr Biochem. 2010 Aug;21(8):717-25. doi: 10.1016/j.jnutbio.2009.04.012. Epub 2009 Jul 18. PMID 19616930
- [Background] Marin M, Maria Giner R, Rios JL, Recio MC. Intestinal anti-inflammatory activity of ellagic acid in the acute and chronic dextrane sulfate sodium models of mice colitis. J Ethnopharmacol. 2013 Dec 12;150(3):925-34. doi: 10.1016/j.jep.2013.09.030. Epub 2013 Oct 17. PMID 24140585
- [Background] Martin DA, Bolling BW. A review of the efficacy of dietary polyphenols in experimental models of inflammatory bowel diseases. Food Funct. 2015 Jun;6(6):1773-86. doi: 10.1039/c5fo00202h. PMID 25986932
- [Background] Mesko B, Poliska S, Szegedi A, Szekanecz Z, Palatka K, Papp M, Nagy L. Peripheral blood gene expression patterns discriminate among chronic inflammatory diseases and healthy controls and identify novel targets. BMC Med Genomics. 2010 May 5;3:15. doi: 10.1186/1755-8794-3-15. PMID 20444268
- [Background] Miller CA, Corbin KD, da Costa KA, Zhang S, Zhao X, Galanko JA, Blevins T, Bennett BJ, O'Connor A, Zeisel SH. Effect of egg ingestion on trimethylamine-N-oxide production in humans: a randomized, controlled, dose-response study. Am J Clin Nutr. 2014 Sep;100(3):778-86. doi: 10.3945/ajcn.114.087692. Epub 2014 Jun 18. PMID 24944063
- [Background] Pellegrini N, Salvatore S, Valtuena S, Bedogni G, Porrini M, Pala V, Del Rio D, Sieri S, Miglio C, Krogh V, Zavaroni I, Brighenti F. Development and validation of a food frequency questionnaire for the assessment of dietary total antioxidant capacity. J Nutr. 2007 Jan;137(1):93-8. doi: 10.1093/jn/137.1.93. PMID 17182807
- [Background] Rosillo MA, Sanchez-Hidalgo M, Cardeno A, de la Lastra CA. Protective effect of ellagic acid, a natural polyphenolic compound, in a murine model of Crohn's disease. Biochem Pharmacol. 2011 Oct 1;82(7):737-45. doi: 10.1016/j.bcp.2011.06.043. Epub 2011 Jul 7. PMID 21763290
- [Background] Rosillo MA, Sanchez-Hidalgo M, Cardeno A, Aparicio-Soto M, Sanchez-Fidalgo S, Villegas I, de la Lastra CA. Dietary supplementation of an ellagic acid-enriched pomegranate extract attenuates chronic colonic inflammation in rats. Pharmacol Res. 2012 Sep;66(3):235-42. doi: 10.1016/j.phrs.2012.05.006. Epub 2012 Jun 4. PMID 22677088
- [Background] Schoepfer AM, Trummler M, Seeholzer P, Seibold-Schmid B, Seibold F. Discriminating IBD from IBS: comparison of the test performance of fecal markers, blood leukocytes, CRP, and IBD antibodies. Inflamm Bowel Dis. 2008 Jan;14(1):32-9. doi: 10.1002/ibd.20275. PMID 17924558
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Snyder SM, Reber JD, Freeman BL, Orgad K, Eggett DL, Parker TL. Controlling for sugar and ascorbic acid, a mixture of flavonoids matching navel oranges significantly increases human postprandial serum antioxidant capacity. Nutr Res. 2011 Jul;31(7):519-26. doi: 10.1016/j.nutres.2011.06.006. PMID 21840468
- [Background] Tibble JA, Sigthorsson G, Bridger S, Fagerhol MK, Bjarnason I. Surrogate markers of intestinal inflammation are predictive of relapse in patients with inflammatory bowel disease. Gastroenterology. 2000 Jul;119(1):15-22. doi: 10.1053/gast.2000.8523. PMID 10889150
- [Background] Valerii MC, Ricci C, Spisni E, Di Silvestro R, De Fazio L, Cavazza E, Lanzini A, Campieri M, Dalpiaz A, Pavan B, Volta U, Dinelli G. Responses of peripheral blood mononucleated cells from non-celiac gluten sensitive patients to various cereal sources. Food Chem. 2015 Jun 1;176:167-74. doi: 10.1016/j.foodchem.2014.12.061. Epub 2014 Dec 23. PMID 25624220
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] Wilson A, Teft WA, Morse BL, Choi YH, Woolsey S, DeGorter MK, Hegele RA, Tirona RG, Kim RB. Trimethylamine-N-oxide: A Novel Biomarker for the Identification of Inflammatory Bowel Disease. Dig Dis Sci. 2015 Dec;60(12):3620-30. doi: 10.1007/s10620-015-3797-3. Epub 2015 Jul 10. PMID 26160437
- [Result] Scaioli E, Belluzzi A, Ricciardiello L, Del Rio D, Rotondo E, Mena P, Derlindati E, Danesi F. Pomegranate juice to reduce fecal calprotectin levels in inflammatory bowel disease patients with a high risk of clinical relapse: Study protocol for a randomized controlled trial. Trials. 2019 Jun 6;20(1):327. doi: 10.1186/s13063-019-3321-8. PMID 31171016
- [Derived] Minato I, Mena P, Ricciardiello L, Scaioli E, Belluzzi A, Rotondo E, Derlindati E, Montanini B, Michelini C, Tosi N, Agullo Garcia V, Picone G, Mengucci C, Dobani S, Salamanca P, Rosi A, Dall'Asta M, Bresciani L, Curti C, Spisni E, Dei Cas A, Bordoni A, Tomas-Barberan FA, Ferguson LR, Del Rio D, Danesi F. Evidence for a Modulatory Effect of a 12-Week Pomegranate Juice Intervention on the Transcriptional Response in Inflammatory Bowel Disease Patients Reducing Fecal Calprotectin Levels: Findings From a Proof-of-Principle Study. Mol Nutr Food Res. 2025 Aug;69(15):e70067. doi: 10.1002/mnfr.70067. Epub 2025 Apr 21. PMID 40255128